CLINICAL TRIAL: NCT02206828
Title: Observational Registry Study for Symbotex™ Composite Mesh in Ventral Hernia Repair
Brief Title: The SymCHro - Observational Registry Study for Symbotex™ Composite Mesh in Ventral Hernia Repair
Acronym: SymCHro
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVSYMB0441
Record Dates: First submitted 2014-07-21; First posted 2014-08-01 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Ventral Incisional Hernia
Keywords: HERNIA; SYMCHRO; SOFRADIM; REGISTRY; SYMBOTEX
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1 GROUP: Only 1 group not predetermined

SUMMARY:
The aim of this Observational Registry Study is to assess the short- and long-term clinical outcomes following the use of Symbotex™ Composite Mesh in primary and incisional abdominal wall hernia surgeries by open or laparoscopic approach, according to the Instruction for use (IFU).

DETAILED DESCRIPTION:
This is an observational multicenter registry study. One hundred consecutive, adult patients scheduled for primary and incisional abdominal wall hernia surgeries using Symbotex™ Composite Mesh will be reported in the ClubHernie online database, with standard data captured of all preoperative, perioperative and post-operative data, for patient's outcomes measurements.

Primary Objective:

Evaluate the incidence of peri-operative and post-operative complications, with postoperative evaluations occurring, at discharge , 1 week (D1 and D8 follow up), 1 month (D30 follow up), 1 year and 2 year follow up after primary and incisional abdominal wall hernia surgeries using Symbotex™ Composite Mesh by open or laparoscopic approach (such as anticipated device related complications such as pain, recurrence, complications related to adhesions, wound complications, other postoperative complications, (SAE).

This online database consists of a systematic and consecutive data entry of all patients treated for Inguinal Hernia and Ventral Hernia by the 30 French surgeon members, with standard data captured of all preoperative, perioperative and post-operative data.

The database is required to be completed anonymously. Quality data control of all data captured into the online database will be performed by coherence analysis by Club Hernie authorized representative;A statistical analysis plan will be developed by Covidien.

Study reported device-related events will be reviewed periodically to assess for any potential trends

ELIGIBILITY:
Inclusion Criteria:

* The first one hundred consecutive adult patients scheduled for primary and incisional abdominal wall hernia surgery by Club Hernie members surgeons using Symbotex™Composite Mesh ;- All patients regardless of gender ≥ 18 years of age presenting with ventral hernias.
* Patients will be informed by surgeon with a written information notice of the nature of the observational registry study.

Exclusion Criteria:

* No exclusion criteria outside the product IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients scheduled for primary and incisional abdominal wall hernia surgeries
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Gillion, Principal Investigator — ICMJE
Locations (1):
- Club Hernie association represented by Dr Gillion, in his capacity as President, Montrouge, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Symbotex Composite Mesh: Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach.
Period: Overall Study
Arm/Group | Symbotex Composite Mesh
Started | 100
Completed | 93
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: 100 patients exhibited ventral hernia
Arm/Group | Symbotex Composite Mesh
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 100

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Peri-operative and Post-operative Complications
Description: Primary endpoint focuses on complications (including recurrence) occurring during procedure, and in short, mid and long-term (measured at 1 month, 1 year and 2 year follow-up respectively) following ventral hernia repair.
  All peri-, intra- and post- operative complications
Time Frame: Various (measured at 1 month, 1 Year & 2 Year)
Population: 6 patients are lost to follow up at 1 year - 7 patients are lost to follow up at 2 year , it is described in the Participant Flow module Outcomes measure reflect Patients who completed each visits
Measure: Count of Participants; unit: Participants
Groups:
- Recurence Rate at 1 Month; Recurrence Rate at 1 Year; Recurrence Rate at 2 Year: Recurrence rate following patients treated for ventral hernia
Arm/Group | Recurence Rate at 1 Month | Recurrence Rate at 1 Year | Recurrence Rate at 2 Year
Number analyzed (Participants) | 100 | 94 | 93
Participants | 0 | 1 | 0

2. Secondary Outcome: Pain Assessment Measured With VAS Score
Description: Pain assessment measured with VAS* score
  *VAS: The postoperative pain is assessed using a 0-10 Visual Analogue Scale. Worst pain experienced over the last 24 hours. Mild pain for VAS score between 0 and 3; Moderate pain for VAS score > 3 and > 6 ; Severe pain for VAS scores > 6
Time Frame: Various ( Baseline Day 0, Day 1, Day 8, Month 1, Month 3, 1 year , 2 year
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- VAS Pain Assessment Day 0: Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
- VAS Pain Assessment Day 1; VAS Pain Assessment Day 8; VAS Pain Assessment Month 1; VAS Pain Assessment Month 3; VAS Pain Assessment 1 Year; VAS Pain Assessment 2 Year: Ease of use Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
Arm/Group | VAS Pain Assessment Day 0 | VAS Pain Assessment Day 1 | VAS Pain Assessment Day 8 | VAS Pain Assessment Month 1 | VAS Pain Assessment Month 3 | VAS Pain Assessment 1 Year | VAS Pain Assessment 2 Year
Number analyzed (Participants) | 82 | 79 | 76 | 79 | 24 | 3 | 2
units on a scale | 4.7 (2.5) | 3.9 (1.8) | 2.0 (1.7) | 0.8 (1.8) | 0.2 (0.7) | 0.0 (0.0) | 0.0 (0.0)

3. Secondary Outcome: Quality of Life for Patient
Description: Quality of Life of patients treated for ventral hernia For long-term follow up, two sets of self-administered Quality of Life (QOL) and patient satisfaction questionnaires were administered by phone call at 1 year and 2 year follow-up.
Time Frame: Various ( 1 Month, 1 year and 2 Year follow up)
Measure: Count of Participants; unit: Participants
Groups:
- Quality of Life at 1 Month; Quality of Life at 1 Year; Quality of Life at 2 Year: Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
Arm/Group | Quality of Life at 1 Month | Quality of Life at 1 Year | Quality of Life at 2 Year
Number analyzed (Participants) | 82 | 94 | 93
Participants
  Does the abdominal wall seem firm?: Yes | 0 | 90 | 91
  Does the abdominal wall seem firm?: No | 0 | 4 | 2
  Does the abdominal wall seem firm?: Not assessed | 82 | 0 | 0
  Do you feel a lump?: Yes | 0 | 7 | 2
  Do you feel a lump?: No | 0 | 87 | 91
  Do you feel a lump?: Not assessed | 82 | 0 | 0
  Do you feel any pain or discomfort?: Yes | 20 | 23 | 12
  Do you feel any pain or discomfort?: No | 62 | 71 | 81
  Do you feel any pain or discomfort?: Not assessed | 0 | 0 | 0
  Reoperation needed?: Yes | 0 | 0 | 1
  Reoperation needed?: No | 82 | 94 | 92
  Reoperation needed?: Not assessed | 0 | 0 | 0

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction For long-term follow up, two sets of self-administered Quality of Life (QOL) and patient satisfaction questionnaires were administered by phone call at 1 year and 2 year follow-up.
Time Frame: Various (1 year and 2 year)
Measure: Count of Participants; unit: Participants
Groups:
- Patient Satisfaction At 1 Year; Patient Satisfaction At 2 Year: Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
Arm/Group | Patient Satisfaction At 1 Year | Patient Satisfaction At 2 Year
Number analyzed (Participants) | 94 | 91
Participants
  Excellent | 10 | 7
  Good | 73 | 79
  Medium | 7 | 3
  Bad | 4 | 2

5. Secondary Outcome: Surgeon Satisfaction (Mesh Handling, Mesh Manipulability, Ease of Use)
Description: Mesh ease of use assessed by surgeons using Symbotex™ Composite Mesh for Patients treated for ventral hernia
Time Frame: Day 0 Baseline
Population: Number of Hernia, some patients exhibits more than 1 hernia (100 patients with 105 ventral hernias) Ease of use: results is based on 100 patients and 105 hernias (100 patients enrolled and having 105 hernias) , However results reported of subjects with missing data or not applicable data respectively;
Measure: Count of Units; unit: Hernia
Units Other Than Participants: Hernia
Groups:
- Ease of Use - Mesh Flexibility: Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
- Ease of Use - Mesh Easy to Trim; Ease of Use - Mesh Easy to Insert; Ease of Use - Mesh Memory Shape; Ease of Use - Minimizing Visceral Attachment Property: Ease of use Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
Arm/Group | Ease of Use - Mesh Flexibility | Ease of Use - Mesh Easy to Trim | Ease of Use - Mesh Easy to Insert | Ease of Use - Mesh Memory Shape | Ease of Use - Minimizing Visceral Attachment Property
Number analyzed (Participants) | 97 | 76 | 97 | 92 | 89
Number analyzed (Hernia) | 102 | 80 | 102 | 96 | 92
Hernia
  Satisfying | 102 | 80 | 102 | 94 | 92
  Unsatisfying | 0 | 0 | 0 | 2 | 0

6. Secondary Outcome: Mesh Handling
Description: ease of use / mesh Handling Mesh ease of use assessed by surgeons using Symbotex™ Composite Mesh for Patients treated for ventral hernia- Participant reflect surgeon who asses the feature of the mesh (for example, 68 surgeons agree that marking eases to place the mesh, 34 surgeons agree that the mesh is conformable to the anatomy etc..
Time Frame: Day 0 Baseline
Measure: Number; unit: participants
Groups:
- Mesh Positioning and Deployment: Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
Arm/Group | Mesh Positioning and Deployment
Number analyzed (Participants) | 100
participants
  Marking eases to place | 68
  conformability to the anatomy is useful | 34
  Absence of direction for positioning is useful | 32
  Prothesis Shape memory eases to place | 53
  Mesh transparency eases to place | 74
  Mesh easy to re-place | 51
  The mesh does not twist during stapling | 43

7. Secondary Outcome: The Use of Symbotex™ Composite Mesh During Surgery Hernia Repair
Description: Surgical technique approach for patients treated for ventral hernia with Symbotex™ Composite Mesh
Time Frame: Baseline Day 0
Measure: Count of Participants; unit: Participants
Groups:
- Surgical Approach: Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
Arm/Group | Surgical Approach
Number analyzed (Participants) | 100
Participants
  Open (Laparotomy) | 20
  Laparoscopy | 77
  Open then Laparoscopy | 3

8. Secondary Outcome: The Use of Symbotex™ Composite Mesh and Surgery Duration
Description: Operative Time (min) for patients treated for ventral hernia
Time Frame: Baseline Day 0
Population: 3 approaches of surgery , thus operative time and hospital stay are provided according to the nature of the surgery the unit of Operative time is in minutes (specify in the title see below) And the unit of hospital stay is in days (speify in the title see below) Missing data on 4 patients.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Operative Time (Min): Symbotex™ Composite Mesh for ventral hernia repair by open or laparoscopic approach
Arm/Group | Operative Time (Min)
Number analyzed (Participants) | 96
minutes
  Open (Laparotomy): number analyzed (Participants) | 19
  Open (Laparotomy) | 67.4 (25.8)
  Laparoscopy: number analyzed (Participants) | 74
  Laparoscopy | 36.2 (23.5)
  Open then Laparoscopy: number analyzed (Participants) | 3
  Open then Laparoscopy | 68.3 (32.1)

9. Secondary Outcome: The Use of Symbotex™ Composite Mesh and Hospital Stay Duration
Description: Hospital stay (Days) for patients treated for ventral hernia with Symbotex Composite mesh device
Time Frame: Baseline Day 0
Population: For 8 patients there is 8 missing data respectively
Measure: Mean (Standard Deviation); unit: days
Groups:
- Hospital Stay ( Days): Hospital stay for patients treated for ventral hernia (Days)
Arm/Group | Hospital Stay ( Days)
Number analyzed (Participants) | 89
days
  Open (Laparotomy): number analyzed (Participants) | 17
  Open (Laparotomy) | 4.7 (2.0)
  Laparoscopy: number analyzed (Participants) | 72
  Laparoscopy | 1.6 (1.6)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Symbotex Composite Mesh
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 9/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbotex Composite Mesh (N=100)
Seroma (Blood and lymphatic system disorders) | 6
Transitory ileus (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-03-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT02206828/Prot_001.pdf
  • Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02206828/SAP_000.pdf